CLINICAL TRIAL: NCT06272773
Title: The Influence of Breathing Pattern on Measurement of Forced Oscillation in Patients With Asthma
Brief Title: Forced Oscillation and Breathing Pattern in Asthma
Status: Not yet recruiting | Type: Observational
Sponsor: Karl Sylvester (Other)
Responsible Party: Sponsor-Investigator, Karl Sylvester, Consultant Healthcare Scientist, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: IRAS Ref: 333663
Record Dates: First submitted 2024-02-16; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Forced Oscillation Test — Participant will breathe normally through the device which sends different frequency sounds into the airways, monitoring the response coming back from central and peripheral airways to calculate airway impedence, reactance and resistance.

SUMMARY:
Asthma is a chronic respiratory disease characterised by airway inflammation, bronchoconstriction, and airway hyperresponsiveness. Accurate and reliable assessment of lung function is crucial in diagnosing and monitoring asthma. The forced oscillation technique (FOT) is a non-invasive method that has gained attention in recent years as a valuable tool for evaluating respiratory mechanics in asthma.

FOT involves applying small amplitude oscillations at various frequencies to the respiratory system and measuring the resulting pressure and flow responses. These measurements provide valuable insights into the mechanical properties of the airways, including resistance, compliance, and reactance. FOT offers several advantages over traditional spirometry, such as its ability to assess peripheral airway function, sensitivity to small airway abnormalities, and ease of use, particularly in young children or individuals with severe airflow limitation. FOT also allows for assessment of respiratory mechanics in individuals who may struggle with performing spirometry manoeuvres.

However, it is unclear whether a change in breathing pattern in patients with obstructive lung disease impacts the assessment of a response to treatment utilising FOT.

Several studies have demonstrated a high prevalence of Breathing Pattern Disorders (BPDs) in individuals with asthma. These findings suggest that BPDs may be common in asthma and could contribute to the manifestation and severity of respiratory symptoms. Evidence suggests that BPDs can adversely affect pulmonary function in individuals with asthma. One study demonstrated that children with asthma and dysfunctional breathing exhibited significantly reduced forced expiratory volume in one second (FEV1) compared to asthmatics without BPD. This suggests that abnormal breathing patterns may contribute to airflow limitation in asthma, leading to decreased lung function.

We therefore wish to determine the impact of different breathing frequencies on parameters measured using FOT in patients diagnosed with asthma and concomitant obstructive lung function abnormality.

DETAILED DESCRIPTION:
Asthma is a chronic respiratory disease characterised by airway inflammation, bronchoconstriction, and airway hyperresponsiveness. Accurate and reliable assessment of lung function is crucial in diagnosing and monitoring asthma. The forced oscillation technique (FOT) is a non-invasive method that has gained attention in recent years as a valuable tool for evaluating respiratory mechanics in asthma.

FOT involves applying small amplitude oscillations at various frequencies to the respiratory system and measuring the resulting pressure and flow responses. These measurements provide valuable insights into the mechanical properties of the airways, including resistance, compliance, and reactance. FOT offers several advantages over traditional spirometry, such as its ability to assess peripheral airway function, sensitivity to small airway abnormalities, and ease of use, particularly in young children or individuals with severe airflow limitation. FOT also allows for assessment of respiratory mechanics in individuals who may struggle with performing spirometry manoeuvres.

Numerous studies have investigated the utility of FOT in diagnosing asthma. For instance, Smith et al. (2018) conducted a study on 100 adults with suspected asthma and found that FOT parameters, such as total respiratory resistance and respiratory system reactance, demonstrated good diagnostic accuracy compared to spirometry. Similarly, Andersson et al. (2020) evaluated the diagnostic performance of FOT in children with asthma and reported that FOT parameters correlated well with markers of airway inflammation, suggesting its potential for identifying asthmatic phenotypes.

In addition to its diagnostic value, FOT has shown promise in monitoring asthma control and assessing treatment response. A study by Van der Wiel et al. (2019) investigated the use of FOT in adults with mild to moderate asthma and found that changes in FOT parameters, such as frequency dependence of resistance and reactance, were sensitive to improvements in lung function following treatment. Similarly, Song et al. (2021) conducted a systematic review and meta-analysis and reported that FOT parameters exhibited significant changes in response to different asthma treatments, supporting its utility as an outcome measure in clinical trials.

However, it is unclear whether a change in breathing pattern in patients with obstructive lung disease impacts the assessment of a response to treatment utilising FOT. Several studies have demonstrated a high prevalence of BPDs in individuals with asthma. In a study by Thomas et al. (2018), 54% of asthma patients exhibited abnormal breathing patterns, characterized by upper chest breathing, reduced diaphragmatic excursion, and increased accessory muscle use. These findings suggest that BPDs may be common in asthma and could contribute to the manifestation and severity of respiratory symptoms. Evidence suggests that BPDs can adversely affect pulmonary function in individuals with asthma. A study by Porges et al. (2019) demonstrated that children with asthma and dysfunctional breathing exhibited significantly reduced forced expiratory volume in one second (FEV1) compared to asthmatics without BPD. This suggests that abnormal breathing patterns may contribute to airflow limitation in asthma, leading to decreased lung function.

Howlett-Foster et al (2022) demonstrated no significant difference in FOT parameters across multiple breathing frequencies in healthy young adults. However, in obstructive lung disease the airway luminal size is smaller due to airway inflammation, excessive smooth muscle contraction and mucus plugging. Based on the Hagen-Poiseuille equation halving the luminal radius increases airways resistance 16-fold. In addition, based on the law of Bernoulli, this smaller luminal size will increase the velocity of air through the airways, reducing airway pressure and leading to a tendency of the airways to narrow further. Therefore, in asthmatic patients a change in breathing frequency may lead to an increase in airway velocity, a reduction in luminal size and hence an increase in airway resistance. A change in breathing pattern between measurements, particularly following treatment administration, may over or underestimate treatment response if the response is measured using FOT and may not be due to the treatment itself.

We therefore wish to determine the impact of different breathing frequencies on parameters measured using FOT in patients diagnosed with asthma and concomitant obstructive lung function abnormality.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18years Confirmed diagnosis of asthma Evidence of obstructive lung disease, FEV1/forced vital capacity (FVC) <lower limit of normal (LLN)

Exclusion Criteria:

* Unstable/Uncontrolled asthma, as designated by the patient's consultant Known breathing pattern disorder Inability to cooperate with instructions Refusal to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with physician-diagnosed asthma and demonstrable obstructive lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in airway resistance at 5 Hertz (Hz) and 19Hz | 20 mins
  To assess the affect of a change in breathing frequency on FOT measurements, specifically airway resistance at 5Hz and 19Hz, in patients with a known diagnosis of asthma.

IPD SHARING:
Plan to Share IPD: Undecided